CLINICAL TRIAL: NCT06292689
Title: A Phase II, Single-arm, Multicenter, Prospective Study of Cardunolizumab in Recurrent or Metastatic Vulvar and Vaginal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: Akeso (Industry); Innovent Biologics, Inc. (Other)
Responsible Party: Principal Investigator, Hanmei Lou, Director, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2024-5(IIT)
Record Dates: First submitted 2024-02-19; First posted 2024-03-05 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Vulvar and Vaginal Cancer
Keywords: Cardunolizumab; Vulvar Cancer; Vaginal Cancer
MeSH Terms: conditions — Vaginal Neoplasms; Vulvar Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): 1.Not systematically treated: 20 patients with recurrent or metastatic vulvar and vaginal cancers enrolled without systemic treatment (platinum-based doublet chemotherapy) will be treated with cardunolizumab + platinum-based doublet chemotherapy ± bevacizumab.
  2.Previous systematic treatment: Twenty patients with recurrent or metastatic vulvar and vaginal cancers previously treated with systemic therapy (platinum-based doublet chemotherapy) will be enrolled as subjects receiving cardunolizumab ± investigator's choice of chemotherapy ± bevacizumab.
  Interventions: Drug: Cardunolizumab

INTERVENTIONS:
Drug: Cardunolizumab — 1. Not systematically treated:
     Cardunolizumab (10mg/kg) + Cisplatinum (50mg/m2)/ Carboplatinum (AUC 4-5) + Paclitaxel (175mg/m2) ± Bevacizumab (15mg/kg) for 6 cycles, every 3 weeks (Q3W), and then Cardunolizumab ± Bevacizumab Q3W maintenance treatment.
  2. Previous systematic treatment:
  Cardunolizumab (10mg/kg) + Chemotherapy regimen selected by the investigator ± Bevacizumab (15mg/kg) for 6 cycles, every 3 weeks (Q3W), and then Cardunolizumab ± Bevacizumab Q3W maintenance treatment.

SUMMARY:
To evaluate the efficacy and safety of cardunolizumab in combination with/without chemotherapy ± bevacizumab for recurrent or metastatic vulvar and vaginal cancers that are not amenable to radical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary enrolment in the study with written informed consent and ability to comply with protocol requirements visits and related procedures as specified in the protocol.
2. Age≥18 & ≤75.
3. Recurrent or metastatic vulvar and vaginal carcinoma not amenable to curative treatment, diagnosed histologically or cytologically, with a pathological type of squamous, adenocarcinoma or adenosquamous carcinoma.
4. Has at least one measurable lesion based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 assessed by investigator. Lesions located in previously irradiated areas are considered measurable if they show progression in such lesions.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Life expectancy of at least 3 months.
7. Prior immunotherapy, targeted therapies are permitted if treatment has not been discontinued due to a grade ≥2 adverse event.
8. The end of prior systemic therapy must be ≥ 4 weeks or 5 half-lives, whichever is shorter, from the first dose of this study. and the treatment-related AE returned to CTCAE 5.0 ≤ Grade 1 (except alopecia and malaise).
9. All participants must provide an archived tumour tissue sample (formalin-fixed paraffin-embedded [FFPE] tissue wax block or a minimum of 5 unstained tumour tissue section samples, preferably newly obtained tumour tissue samples) within 2 years prior to randomisation.
10. Has adequate organ function.
11. Have agreed to take effective contraception from the date of signing the informed consent form until 120 days after the last administration.
12. Ability to understand and sign written informed consent and to comply with programme visits and related procedures.

Exclusion Criteria:

1. Participants who have received prior systemic anticancer therapy (including study drug) within 4 weeks prior to the first dose of study treatment. Note: If participants have undergone major surgery, they must have fully recovered from the toxicity and/or complications of the treatment prior to starting study treatment. Patients who require elective major surgical treatment during the study period are not eligible for enrolment.
2. Participants must have recovered to grade ≤1 or baseline level from all AEs resulting from prior treatment.
3. Received radiotherapy within 2 weeks prior to the first dose. For patients who have received radiotherapy prior to 2 weeks before the first dose, all of the following conditions must be met for enrolment: glucocorticosteroids are not required, and radiation pneumonitis, radiation hepatitis, and radiation enteritis are excluded. Patients with palliative radiotherapy to bone lesions more than 7 days from the first dose may be enrolled. Reirradiation of previously treated sites is not permitted.
4. Received an immunomodulatory drug within 2 weeks prior to randomisation.
5. Active Hepatitis B or Hepatitis C.
6. History of severe bleeding tendency or coagulation disorder.
7. Pregnant or lactating female patients.
8. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of this subject to participate, in the opinion of the treating investigator.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2026-03-22 (Estimated); Study Completion 2027-03-22 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 2 years
  ORR is defined as the proportion of subjects with confirmed CR or PR, based on RECIST v1.1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 2 years
  PFS is defined as the time from the start of treatment with Cardunolizumab until the first documentation of disease progression or death due to any cause, whichever occurs first.
Overall survival (OS) | Up to 2 years
  OS is defined as the time from the start of treatment with Cardunolizumab until death due to any cause.
Disease control rate (DCR) | Up to 2 years
  DCR is defined as the proportion of subjects with confirmed CR, PR, or SD, based on RECIST v1.1.
Duration of response (DOR) | Up to 2 years
  DOR is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
Adverse events (AEs) | From first dose of Cardunolizumab through to 90 days after last dose of Cardunolizumab
  Incidences of treatment-emergent adverse events (TEAEs) , treatment-related adverse events (TRAEs) as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China